CLINICAL TRIAL: NCT06686160
Title: Comparative Effects of Plyometric Training and Theraband Resistant Exercises on Agility, Power and Dynamic Balance in Karate Players With Patello Femoral Pain Syndrome
Brief Title: Comparative Effects of Plyometric Training and Theraband Resistant Exercises in Karate Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0411
Record Dates: First submitted 2024-10-24; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Sports Physical Therapy
Keywords: Muscle imbalance; Patellofemoral pain; Theraband Resistance exercises
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training (Experimental): Patient will be given baseline treatment that includes thermotherapy+ TENS+ low intensity high repetition exercises. After we will apply our basic intervention exercise, Plyometrics are primarily used by athletes to improve performance and are used in the fitness field to a much lesser degree. This training focuses on learning to move from a muscle extension to a contraction in a explosive way, for example repeated jumping.
  Interventions: Other: Plyometrics Training
- Theraband Resistance Exercise (Experimental): Patient will be given baseline treatment that includes thermotherapy+ TENS+ low intensity high repetition exercises. After we will apply our basic intervention exercise Therabands is a Set of bands which are primarily use for resistance Training for strength and Power.
  Interventions: Other: Theraband Resistance Exercise

INTERVENTIONS:
Other: Plyometrics Training — Patient will be given baseline treatment that includes thermotherapy+ TENS+ low intensity high repetition exercises. After we will apply our basic intervention exercise, Plyometrics are primarily used by athletes to improve performance and are used in the fitness field to a much lesser degree. This training focuses on learning to move from a muscle extension to a contraction in a explosive way, for example repeated jumping.
  Arms: Plyometric Training
Other: Theraband Resistance Exercise — Patient will be given baseline treatment that includes thermotherapy+ TENS+ low intensity high repetition exercises. After we will apply our basic intervention exercise Therabands is a Set of bands which are primarily use for resistance Training for strength and Power.
  Arms: Theraband Resistance Exercise

SUMMARY:
The aim of this study is to find out the Comparative effects of Plyometric training and Theraband Resistant Exercises on Agility, Power and Dynamic balance in karate Players with Patellofemoral Syndrome. Understanding how these methods impact agility, power, and dynamic balance provides practical insights for designing rehabilitation programs.It help therapists to find which evidence-based recommendations are beneficial for maximizing the athletes agility, power, dynamic balance and overall performance or well-being of the karate players with Patellofemoral pain syndrome.

DETAILED DESCRIPTION:
The literature gap in this study on the Comparative Effects of Plyometric Training and Theraband Resistant Exercises on Agility, Power and Dynamic Balance in Karate Players with Patellofemoral Syndrome may exist, there might be limited studies specifically addressing this unique combination of factors, further investigation is needed to explore the evidence based effect of these exercises on karate players with Patellofemoral syndrome, considering the interplay between the exercises and the sport specific demands.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age 18 to 25 years
* With playing experience of 3 to 5 years will be included
* Minimum Sports activity 1 hour 4 times a week
* Positive patella femoral compression test (Pain is in around the patella and back of knee cap)

Exclusion Criteria:

* Recreational players
* Players with recent injury in past 6 months
* Any musculoskeletal and neurological problem
* Player addicted to any drug or alcohol will be excluded

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 weeks
  Numeric Pain Rating Scale NPRS is based on 11-point numerical rating scale for determining pain intensity, 0(no pain) to 10(worst pain imaginable) pain intensity .NRS pain has high validity and reliability (β = 0.42 [95% CI 0.04, 0.80]
The Kujalapatello femoral | 6 weeks
  The Kujalapatellofemoral score is one of the commonly used assessment scales for patients with PFP. It provides a functional assessment instrument for knee complaints related to the patellofemoral structure. The scale was designed especially for patients withscoring system will be perform to diagnose Patello femoral syndrome,with a variable ordinal response format high internal consistency (αCoef = 0.83 to 0.91)
Agility T Test | 6 weeks
  Agility will be measured by the agility T-tests,high intra-trail reliability of the test (ICC=0.98). The participants were instructed to run 9.14 meters from the starting line to the first cone, touch the tip with their right hand, shuffle 4.57 meters to the left to the second cone, shuffle 9.14 meters to the right to the third cone, touch with their right hand, shuffle 4.57 meters to the left to the middle cone, touch with their left hand, and then backpedal to the starting line.
Star Excursion Balance Test | 6 weeks
  The Star Excursion Balance Test (SEBT) is a dynamic test that requires strength, flexibility, and proprioception Star Excursion Balance Test (SEBT) the intra class correlation coefficients ( 0.86 to 0.92).The SEBT is performed with the subject standing at the center of a grid placed on the floor, with 8 lines extending at 45° increments from the center of the grid. The 8 lines positioned on the grid are labeled according to the direction of excursion relative to the stance leg. The plane was constructed in a facility with the help of a protractor and adhesive tape on the hard tile floor.
40-Yd Speed Test | 6 weeks
  Speed will be measured by the 40-Yd Sprint Test. The test involves running a single maximum sprint over 40 yards, with the time recorded. The aim of this test will be to determine 40-Yd Sprint. Sprints of 40 yd were used to determine quickness ICC > 0.987.
Sargent Test | 6 weeks
  To mark the wall at the height of their jump, the participant applies chalk to the tips of their fingers. After standing away from the wall, the individual uses both arms and legs to help project their body upwards and jumps as high as they can. At the peak of the jump, they try to make contact with the wall. Power will be measured by the Sargent Test. Vertical Jump test is a very common test for measuring explosive leg power intra-rater class reliability ICC = 0.903 to 0.934.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Muaaz, DPT, Principal Investigator — Riphah International University
Locations (1):
- Youth karate Acadmy, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willy RW, Hoglund LT, Barton CJ, Bolgla LA, Scalzitti DA, Logerstedt DS, Lynch AD, Snyder-Mackler L, McDonough CM. Patellofemoral Pain. J Orthop Sports Phys Ther. 2019 Sep;49(9):CPG1-CPG95. doi: 10.2519/jospt.2019.0302. PMID 31475628
- [Background] Sisk D, Fredericson M. Update of Risk Factors, Diagnosis, and Management of Patellofemoral Pain. Curr Rev Musculoskelet Med. 2019 Dec;12(4):534-541. doi: 10.1007/s12178-019-09593-z. PMID 31773479
- [Background] Lee JH, Jang KM, Kim E, Rhim HC, Kim HD. Static and Dynamic Quadriceps Stretching Exercises in Patients With Patellofemoral Pain: A Randomized Controlled Trial. Sports Health. 2021 Sep-Oct;13(5):482-489. doi: 10.1177/1941738121993777. Epub 2021 Feb 20. PMID 33615901
- [Background] Lee JH, Shin KH, Han SB, Sun Hwang K, Lee SJ, Jang KM. Prospective comparative study between knee alignment-oriented static and dynamic balance exercise in patellofemoral pain syndrome patients with dynamic knee valgus. Medicine (Baltimore). 2022 Sep 16;101(37):e30631. doi: 10.1097/MD.0000000000030631. PMID 36123932
- [Background] Gaitonde DY, Ericksen A, Robbins RC. Patellofemoral Pain Syndrome. Am Fam Physician. 2019 Jan 15;99(2):88-94. PMID 30633480
- [Background] Fick CN, Jimenez-Silva R, Sheehan FT, Grant C. Patellofemoral kinematics in patellofemoral pain syndrome: The influence of demographic factors. J Biomech. 2022 Jan;130:110819. doi: 10.1016/j.jbiomech.2021.110819. Epub 2021 Oct 15. PMID 34749164
- [Background] Zambarano EK, Bazett-Jones DM, de Oliveira Silva D, Barton CJ, Glaviano NR. Confidence and Knowledge of Athletic Trainers in Managing Patellofemoral Pain. J Athl Train. 2022 Jan 1;57(1):79-91. doi: 10.4085/1062-6050-0279.21. PMID 35040987
- [Background] Neal BS, Lack SD, Lankhorst NE, Raye A, Morrissey D, van Middelkoop M. Risk factors for patellofemoral pain: a systematic review and meta-analysis. Br J Sports Med. 2019 Mar;53(5):270-281. doi: 10.1136/bjsports-2017-098890. Epub 2018 Sep 21. PMID 30242107
- [Background] Emamvirdi M, Letafatkar A, Khaleghi Tazji M. The Effect of Valgus Control Instruction Exercises on Pain, Strength, and Functionality in Active Females With Patellofemoral Pain Syndrome. Sports Health. 2019 May/Jun;11(3):223-237. doi: 10.1177/1941738119837622. Epub 2019 Apr 29. PMID 31034336
- [Background] Saad MC, Vasconcelos RA, Mancinelli LVO, Munno MSB, Liporaci RF, Grossi DB. Is hip strengthening the best treatment option for females with patellofemoral pain? A randomized controlled trial of three different types of exercises. Braz J Phys Ther. 2018 Sep-Oct;22(5):408-416. doi: 10.1016/j.bjpt.2018.03.009. Epub 2018 Apr 4. PMID 29661570
- [Background] Tramontano M, Pagnotta S, Lunghi C, Manzo C, Manzo F, Consolo S, Manzo V. Assessment and Management of Somatic Dysfunctions in Patients With Patellofemoral Pain Syndrome. J Am Osteopath Assoc. 2020 Mar 1;120(3):165-173. doi: 10.7556/jaoa.2020.029. PMID 32091560
- [Background] Kasitinon D, Li WX, Wang EXS, Fredericson M. Physical Examination and Patellofemoral Pain Syndrome: an Updated Review. Curr Rev Musculoskelet Med. 2021 Dec;14(6):406-412. doi: 10.1007/s12178-021-09730-7. Epub 2021 Oct 29. PMID 34713383